CLINICAL TRIAL: NCT06131749
Title: Genital Tract Infections, the Vaginal Microbiome and Gestational Age at Birth Among Pregnant Women in South Africa
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Foundation for Professional Development (Unknown); Utrecht University (Other); University of Pretoria (Other); University of Cape Town (Other); University of Southern California (Other); University of Alabama at Birmingham (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Other Study IDs: SNSF197831
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sexually Transmitted Infections (Not HIV or Hepatitis); Premature Birth; Pregnancy; Infection; Microbial Colonization; Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection; Trichomonas Vaginitis; Mycoplasma Genitalium Infection; Bacterial Vaginosis; Vaginal Candida; Ureaplasma Urealyticum Infection; Genital Mycoplasma Infection; HIV Infections
Keywords: Sexually transmitted infections; Preterm birth; Gestational age at birth; Vaginal microbiome; Genital mycoplasmas; Organism load; Vaginal yeast; Antenatal care
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis; Premature Birth; Pregnancy Complications, Infectious; Communicable Diseases; Gonorrhea; Trichomonas Vaginitis; Vaginosis, Bacterial; Candidiasis, Vulvovaginal; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swabs for on-site testing for Chlamydia trachomatis, Neisseria gonorrhoeae. Swabs discarded after testing Vaginal swabs for PCR detection of Trichomonas vaginalis, Candida spp., Mycoplasma genitalium, Mycoplasma hominis, Ureaplasma urealyticum, Ureaplasma parvum. Extracted DNA retained after testing Vaginal specimens for microscopy and Nugent scoring. Specimens retained Vaginal swab for 16S ribosomal ribonucleic acid (rRNA) amplicon sequencing. Extracted DNA retained after testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: No intervention. Followed during pregnancy at baseline and 30-34 weeks. Followed after delivery at 3-6 days.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, observational cohort study

SUMMARY:
This cohort study plans to investigate associations between the presence of multiple lower genital tract microorganisms in pregnancy and gestational age at birth.

The study enrols pregnant women at one public health care facility in East London, South Africa. At enrolment and 30-34 weeks of pregnancy, participants provide swabs for testing for sexually transmitted infections, vaginal yeasts and genital mycoplasmas; for microscopy and Nugent scoring; and for 16S ribosomal ribonucleic acid gene sequencing and quantification. The primary outcome is gestational age at birth.

Statistical analyses include: regression modelling to explore associations between specific microorganisms (including microbiota) and gestational age at birth; construction of an index of vaginal inflammation, using data about microorganism load and inflammatory potential; classification and regression tree analysis to examine which combinations of microorganisms contribute to earlier gestational age at birth.

DETAILED DESCRIPTION:
Background: Preterm birth complications are the most common cause of death in children under 5 years. In South Africa, the prevalence of both genital tract infections and adverse pregnancy outcomes are high. This study takes a holistic approach, investigating both the presence and quantity of multiple lower genital tract microorganisms, including vaginal microbiota, in pregnancy and their associations with gestational age at birth. Specific objectives are to explore: (1) the association between the presence of specific lower genital tract microorganisms and gestational age at birth (primary outcome), as well as secondary adverse pregnancy outcomes; (2) the association between quantified load of vaginal and sexually transmitted microorganisms and gestational age at birth (primary outcome) as well as secondary adverse pregnancy outcomes; and (3) the combinations of microorganisms that are most strongly associated with earlier gestational age at birth.

Methods: This prospective closed cohort study follows women enrolled during pregnancy until after they give birth. This cohort study is part of a larger project, called Philani Ndiphile (meaning 'be healthy and I will be healthy' in isiXhosa).

A trained study field worker checks for eligibility and obtains written informed consent. A study nurse performs an abdominal ultrasound to estimate the gestational age and confirm eligibility.

At the enrolment visit and a follow-up visit at 30-34 weeks, a study nurse collects vaginal specimens for: on-site testing for Chlamydia trachomatis and Neisseria gonorrhoeae (with antibiotic treatment if positive); and offsite testing for: Nugent scoring; detection and quantification of Mycoplasma genitalium, M. hominis, Ureaplasma. parvum, U. Urealyticum, Trichomonas vaginalis, Candida spp. and 16S rRNA amplicon sequencing for vaginal microbiota analyses.

At a post-natal visit, 3-6 days after giving birth, a study nurse collects information about the birth outcome.

Statistical analyses include:

Objective 1. a) univariable and multivariable regression analyses for associations between specific microorganisms and gestational age at birth. b) compositional multivariable analysis methods to analyse individual taxon relative abundances and mixed effects models to assess associations between pregnancy outcome and vaginal microbiota diversity, vaginal microbiota types and absolute abundances of predefined bacterial groups.

Objective 2. Development of a 'vaginal inflammation index', based on quantification of the vaginal microbiota and their inflammatory potential. This vaginal inflammation index will be analysed as a fixed effect in mixed effects models with pregnancy outcomes.

Objective 3. Classification and regression tree analyses to examine the combination of microorganisms that best predicts earlier gestational age at birth.

ELIGIBILITY:
Inclusion Criteria:

* Living in Buffalo City Metropolitan Municipality
* Intend to deliver in the same municipality
* <27 weeks of gestation at enrolment, confirmed by ultrasound
* Provide written informed consent

Exclusion Criteria:

* Participation in any other research study
* Inability to understand and speak a local language (English, Afrikaans, or isiXhosa).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women receiving antenatal care at one primary health care facility in Buffalo City Metropolitan Municipality, Eastern Cape Province, South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth | Recorded within 2 weeks of delivery
  Gestational age in days, estimated using data from obstetric ultrasound at enrolment visit

SECONDARY OUTCOMES:
Preterm birth | Recorded within 2 weeks of birth
  Number of babies liveborn before 37 completed weeks of pregnancy, estimated using data from obstetric ultrasound at enrolment visit
Low birth weight | Measured within 72 hours of birth
  Number of babies with birth weight <2500g
Miscarriage | Collected throughout pregnancy until delivery
  Number of foetuses delivered dead before 28 completed weeks of pregnancy or with birth weight below 1000g. Gestational age estimated using data from obstetric ultrasound at enrolment visit
Stillbirth | Collected throughout pregnancy until delivery
  Number of foetuses delivered dead at or after 28 completed weeks of pregnancy or with birth weight above 1000g at delivery. Gestational age estimated using data from obstetric ultrasound at enrolment visit

OTHER OUTCOMES:
Prevalence of microorganisms | Measured at enrolment visit and at 30-34 week visit
  Number of women with a specific microorganism / number of women tested
Incidence of microorganisms | Measured at 30-34 week visit
  Number of women with new detection of a specific microorganism per 1000 woman years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Low, MD, Principal Investigator — University of Bern
Locations (1):
- Empilweni Gompo Community Health Centre, East London, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gigi RMS, Mdingi MM, Jung H, Claassen-Weitz S, Butikofer L, Klausner JD, Muzny CA, Taylor CM, van de Wijgert JHHM, Peters RPH, Low N. Genital tract infections, the vaginal microbiome and gestational age at birth among pregnant women in South Africa: a cohort study protocol. BMJ Open. 2023 Dec 28;13(12):e081562. doi: 10.1136/bmjopen-2023-081562. PMID 38154893